CLINICAL TRIAL: NCT07319624
Title: Bedside PEEP Selection in by Electrical Impedence Tomography During Mechanical Ventilation in Children
Acronym: BePeSEIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Papa Giovanni XXIII Hospital (Other)
Responsible Party: Principal Investigator, Alfio Bronco, Principal Investigator - Consultant Pediatric Intensivist, Papa Giovanni XXIII Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PETI
Record Dates: First submitted 2025-11-23; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Pneumonia; Tetralogy of Fallot Correction; Caustics Ingestion; Orthotopic Liver Transplantation
Keywords: EIT; PEEP; Mechanical Ventilation; Electrical Impedence Tomography; PARDS
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric Acute Respiratory Distress Syndrome (PARDS) patients (Experimental): Patients under 3 years of age who required mechanical ventilation due to impaired oxygenation or altered respiratory mechanics.
  Interventions: Diagnostic Test: Electrical Impedence Tomography

INTERVENTIONS:
Diagnostic Test: Electrical Impedence Tomography — An EIT belt with 16 electrodes (PulmoVista® 500, Dräger Medical GmbH, Lübeck, Germany) appropriate to the children's weight was placed at the fourth or fifth intercostal space along the axillary line.

SUMMARY:
This prospective study evaluates the feasibility and safety of using Electrical Impedance Tomography (EIT) to guide PEEP selection in mechanically ventilated infants and toddlers under 3 years of age. This population is challenging for its variety and anatomophysiologic peculiarity. A decremental PEEP trial using 1 cmH₂O steps following a recruitment maneuver at 35 cmH₂O was compared between EIT and other best PEEP assessment protocols.

DETAILED DESCRIPTION:
The study enrolled consecutive patients under 3 years of age who required mechanical ventilation due to impaired oxygenation or altered respiratory mechanics. Impaired oxygenation sufficient for inclusion was defined as an oxygenation index (OI) greater than 4, defined as mean airway pressure multiplied by FiO₂ divided by PaO₂, and/or an oxygen saturation index (OSI), defined as mean airway pressure multiplied by FiO₂ divided by SpO₂, greater than 5. Altered respiratory mechanics sufficient for inclusion was defined as reduced respiratory system compliance normalized to body weight (Crs/kg) below 0.7 mL/cmH₂O/kg.

Patients were excluded if they had contraindications to the placement of the EIT belt, such as thoracic fractures, chest drains, or subcutaneous thoracic devices. The presence of intracardiac shunts was also an exclusion criterion. Further exclusions included confirmed or suspected pneumothorax on chest X-ray or lung ultrasound, hemodynamic instability requiring adrenaline or noradrenaline at doses exceeding 0.05 mcg/kg/min, or a reduction in systolic blood pressure greater than 30% during recruitment maneuvers. Technical issues that prevented reliable acquisition of EIT signals, including prolonged signal instability, belt-to-chest size incompatibility (< 3 kg), or the need for urgent clinical interventions, also led to exclusion. Lack of informed consent from parents or legal guardians precluded enrollment.

Study Protocol The stepwise PEEP titration protocol used in this study is partially part of a clinical approach routinely adopted in the PICU of our institution to optimize lung recruitment and individualize ventilator settings in mechanically ventilated children.

According this study protocol, once clinical stabilization was achieved - defined as adequate sedation and analgesia, cardiovascular stability, and appropriate patient-ventilator synchrony -neuromuscular blockade was administered. An EIT belt with 16 electrodes (PulmoVista® 500, Dräger Medical GmbH, Lübeck, Germany) appropriate to the patient's weight was placed at the fourth or fifth intercostal space along the axillary line.

Baseline parameters were collected, including gas exchange data, respiratory mechanics, and ventilator settings (PEEP, tidal volume [Vt], respiratory rate, driving pressure [ΔP], compliance [Crs], FiO₂, SpO₂, OI or OSI), as well as blood gas analysis when available. PEEP was initially set according to the ARDSNet lower PEEP/higher FiO₂ table, referred to as PEEPnih. If children was volume-controlled ventilate, pressure-controlled ventilation was applied with an inspiratory pressure above PEEP equal to the baseline ΔP to maintain a similar Vt regardless of the previous ventilation mode.

A 5-minute EIT baseline recording was performed before initiating the recruitment maneuver.

The maneuver consisted of a sustained inflation at 35 cmH₂O, which was maintained until the global impedance curve displayed a plateau - suggestive of the end of a significant recruitment - or for a maximum duration of 25 seconds. This approach was introduced as a safety measure to avoid unnecessary overdistension and excessive intrathoracic pressures with potential hemodynamic impairment. The use of the impedance-time curve to guide the termination of the sustained inflation is consistent with the method described by Costa et al., which supports the identification of lung recruitment plateau using EIT-derived global impedance monitoring.

Following the recruitment maneuver, a decremental PEEP trial was conducted with 5-minute steps, starting from PEEPnih+4 cmH₂O and progressively decreasing by 1 cmH₂O increments down to PEEPnih-4 cmH₂O. The trial was discontinued early if the global ΔEELI signal dropped by more than 15%, indicating relevant decrease of the end-expiratory lung volume. The trial was also interrupted if clinical concerns arose, such as newly suspected pneumothorax or hemodynamic instability.

At each PEEP step, the following variables were recorded: heart rate, blood pressure, SpO₂, OSI, plateau pressure, ΔP, Vt, global Crs, and the percentage distribution of ventilation in the four ventral to dorsal regions of interest (ROIs). From these, compliance values for gravity-dependant (CrsD - dorsal regions) and non gravity-dependant (CrsND - ventral regions) regions were derived.

ELIGIBILITY:
Inclusion Criteria:

* Age under 3
* Impaired oxygenation - defined as an

  1. oxygenation Index (OI = mean airway pressure multiplied by FiO₂ divided by PaO₂) greater than 4; and/or
  2. an Oxygen Saturation Index (OSI = mean airway pressure multiplied by FiO₂ divided by SpO₂) greater than 5; or
  3. altered respiratory mechanics - defined as reduced respiratory system compliance normalized to body weight (Crs/kg) below 0.7 mL/cmH₂O/kg.

Exclusion Criteria:

* thoracic fractures
* chest drains
* subcutaneous thoracic devices
* presence of intracardiac shunts
* confirmed or suspected pneumothorax on chest X-ray or lung ultrasound
* hemodynamic instability requiring adrenaline or noradrenaline at doses exceeding 0.05 mcg/kg/min, or a reduction in systolic blood pressure greater than 30% during recruitment maneuvers.
* technical issues that prevented reliable acquisition of EIT signals, including prolonged signal instability
* belt-to-chest size incompatibility (< 3 kg)
* lack of informed consent

Ages: 0 Years to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Feasibility (% of patients that complete the EIT-guided PEEP trial) | 20 weeks
  assessing the feasibility of an individualized PEEP titration using an EIT-guided decremental PEEP trial specifically designed for smaller children.

SECONDARY OUTCOMES:
To compare PEEPeit (cmH2O) with PEEPnih (cmH2O) | 20 weeks
  To compare PEEP levels determined by EIT (PEEPeit, cmH2O) with those recommended by NIH tables (PEEPnih, cmH2O) and those identified through the highest static compliance measurements (Compliance-guided method; PEEPCrs, cmH2O)
To evaluate changes of EIT patterns of overdistension (%) and derecruitment (%) according to changes in respiratory system Compliance-guided method (mL/cmH2O) | 20 weeks
  To evaluate changes of EIT patterns of overdistension (%) and derecruitment (%) according to changes in respiratory system Compliance-guided method (mL/cmH2O)
To assess changes in respiratory system compliance (mL/cmH2O) across different PEEP levels (cmH2O) | 20 weeks
  To assess changes in respiratory system compliance (mL/cmH2O) across different PEEP levels (cmH2O)
To assess changes in end-expiratory lung impedance (arbitrary units) by EIT across different PEEP levels (cmH2O) | 20 weeks
  To assess changes in end-expiratory lung impedance (arbitrary units) by EIT across different PEEP levels (cmH2O)
To assess changes in oxygenation (PaO2/FiO2, mmHg) across different PEEP levels | 20 weeks
  To assess changes in oxygenation (PaO2/FiO2, mmHg) across different PEEP levels

CONTACTS AND LOCATIONS:
Overall Officials: Alfio Bronco, MD, Principal Investigator — Papa Giovanni XXIII Hospital, Bergamo, BG 24100
Locations (1):
- Papa Giovanni XXIII Hospital, Bergamo, BG 24100, Bergamo, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Pediatric population sensitive data